CLINICAL TRIAL: NCT01283789
Title: Phase II Trial of Lapatinib and RAD-001 for HER2 Positive Metastatic Breast Cancer
Brief Title: Lapatinib and RAD-001 for HER2 Positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Novartis (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12418
Record Dates: First submitted 2011-01-10; First posted 2011-01-26 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Metastatic Breast Cancer
Keywords: breast; cancer; metastatic; metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Lapatinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib and RAD-001 (Experimental): RAD-001 will be administered orally as a once-daily dose of 5 mg (one 5 mg tablet) continuously from study day 1 until progression of disease or unacceptable toxicity. Patients will be instructed to take RAD-001 in the morning, at the same time each day.
  Lapatinib will be administered orally as a once-daily dose of 1250 mg (five 250 mg tablets) continuously from study day 1 until progression of disease or unacceptable toxicity. Patients will be instructed to take lapatinib at bedtime, at the same time each day. Lapatinib should be taken by the patient in a fasting state.
  Interventions: Drug: Lapatinib and RAD-001

INTERVENTIONS:
Drug: Lapatinib and RAD-001 — Lapatinib will be taken orally as a once-daily dose of 1250 mg (five 250 mg tablets) continuously from study day 1 until progression of disease. Patients will take the tablet at bedtime, at the same time each day, in a fasting state.
  Everolimus will be taken orally as a once-daily dose of 5 mg (one 5 mg tablet) from study day 1 until progression of disease. Patients will take the tablet at the same time each morning.
  Other Names: everolimus; tykerb

SUMMARY:
By doing this study, researchers hope to learn the effectiveness of the combination of Lapatinib and RAD-001 for treating patients who have progressed on previous therapies.

DETAILED DESCRIPTION:
Twenty to twenty five percent of Human Breast Cancers are HER2 positive. HER2 positivity confers a poor prognosis in the absence of HER2 targeted therapies (trastuzumab and lapatinib). With these targeted agents often combined with chemotherapy, the treatment of HER2 positive breast cancer has improved greatly, both in metastatic and adjuvant settings. However most patients with metastatic HER2 positive breast cancer will eventually develop resistance to these agents and succumb to their disease. Therefore, there is a need to test new agents and new combinations that can increase the efficacy of HER2 targeted therapy and/or prevent resistance to HER2 targeted therapies.

A unique feature of HER2 positive breast cancers is a rather high incidence of brain metastasis in this population. Brain metastases develop in one third to one half of patients with advanced HER2+ breast cancer and CNS is a frequent site of trastuzumab failure. Effective therapy for patients with central nervous system (CNS) progression after cranial radiation is extremely limited and represents a major clinical challenge. Compared to trastuzumab, which has no CNS activity, lapatinib, an epidermal growth factor receptor/HER2 inhibitor, has modest CNS activity. In a study of more than 200 patients by Lin et al, 21% of patients experienced a 20% volumetric reduction in their CNS lesions on lapatinib. An association was observed between volumetric reduction and improvement in progression-free survival and neurologic signs and symptoms. Of the 50 evaluable patients who entered the lapatinib plus capecitabine extension, 20% experienced a CNS objective response and 40% experienced a 20% volumetric reduction in their CNS lesions. Mammalian target of Rapamycin (mTOR) is a serine/threonine kinase that regulates key functions associated with cell growth, survival and angiogenesis. mTOR is activated by HER signaling, PI3K oncogenic mutation and loss of PTEN function. In vitro data suggests that activation of mTOR by PTEN loss and PI3K mutation induces trastuzumab resistance. Preclinical studies have shown that mTOR inhibition enhances the efficacy of trastuzumab and reverses trastuzumab resistance caused by PTEN loss. This preclinical finding was confirmed in 2 recent Phase 1 studies where addition of mTOR inhibitor (RAD-001) to trastuzumab and chemotherapy reversed the resistance to Trastuzumab in patients with heavily pretreated metastatic HER2 positive breast cancer. Thus, mTOR inhibition would be an attractive modality to add to HER2 targeted therapy for improving outcomes in women with HER2 positive breast cancer. Everolimus (RAD001), a rapamycin analogue, is an orally administered inhibitor of mTOR. Everolimus has shown promising activity in solid tumors. PK data in mouse models indicated that penetration of rapamycin and Everolimus into the CNS is substantial. Everolimus brain levels are approximately one-third that of systemic levels at 48 hours after a dose.

A small molecule inhibitor of HER2, lapatinib is clinically active in women with advanced HER2-positive breast cancer who have progressed on trastuzumab treatment. However, the effectiveness of this class of agents is limited by either primary resistance or acquired resistance. Using an unbiased genetic approach, Eichhorn et al performed a genome wide loss-of-function short hairpin RNA screen to identify novel modulators of resistance to lapatinib. Tumor suppressor PTEN was identified as a modulator of lapatinib sensitivity in vitro and in vivo. In addition, they show that two dominant activating mutations in PI3K pathway which are prevalent in breast cancer, also confer resistance to lapatinib. They also showed that PI3K-induced lapatinib resistance could be abrogated through the use of NVP-BEZ235, a dual inhibitor of PI3K/mTOR. This suggests that deregulation of the PI3K pathway leads to lapatinib resistance, which can be effectively reversed by inhibition of PI3K/mTOR pathway.

In summary, the combination of Everolimus and lapatinib needs to be studied in women with metastatic breast cancer who have progressed on at least one prior anti-HER2 therapy. If RAD-001 is able to overcome resistance to anti-HER2 therapies, a very desirable response rate and prolongation in TTP can be expected. Moreover, both lapatinib and Everolimus appear to be able to cross the blood brain barrier, and this combination may prove to be effective in controling CNS metastases in this population. The investigators hypothesize that combining mTOR inhibitor Everolimus with lapatinib will be an effective strategy for patients who have progressed on a prior anti-HER2 therapy, both systemically and within the CNS.

ELIGIBILITY:
INCLUSION CRITERIA

* Females > 18 years of age
* Histologically proven adenocarcinoma of breast in primary or metastatic setting. Stage: Locally advanced (inoperable) or metastatic
* HER2 positive breast cancer (IHC 3+ or FISH ratio of > 2.0)
* ECOG Performance status 0-2
* Up to four prior chemotherapy regimens and anti-HER2 agents in metastatic setting allowed. Must have progressed on at least one HER2 targeted therapy (lapatinib or Herceptin) for metastatic breast cancer.
* Women of childbearing potential must have negative urine or serum pregnancy test within 7 days prior to administration of Everolimus. If barrier contraceptives are used, they must be continued throughout trial by both sexes. Hormonal contraceptives not acceptable as a sole method of contraception.
* Adequate kidney function: serum creatinine of < 1.5 mg/dl and/or creatinine clearance of > 60 mL/min
* Adequate hepatic function: transaminases < 2.5 x upper limit of normal (up to 5 x ULN in patients with liver metastases) and total bilirubin < 1.5 mg/dL. Adequate coagulation: INR ≤ 2.0 and PTT < 1.5 X the upper limit of institution normal range. Oral anticoagulants, eg, warfarin are CYP2C9 substrates and, as such, no interaction with Everolimus is expected. Anticoagulation with Coumadin is allowed if target INR is ≤ 2.0 and stable for > 2weeks. Anticoagulation with LMW is allowed.
* Must be informed of investigational nature of study, and must sign an informed consent
* Pretreatment lab values (must be performed within 14 days of patient registration unless otherwise specified. Other baseline studies must be performed within 30 days of registration.
* Patients will have baseline CT chest, abdomen and pelvis within 30 days of registration.
* Adequate cardiac function (LVEF ≥ 50% as measured by echocardiogram or MUGA scan).
* Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, patient may be included after initiation of appropriate lipid lowering medication with approval from the principal investigator.
* Must have measurable or non-measurable disease by RECIST criteria (version 1.1), with radiologic scans performed within 30 days of registration. Baseline scans can include:

  * CT Scan or MRI and Bone Scan OR
  * PET/CT provided it is performed with both IV and oral contrast and the CT is acquired with 5mm or less slice thickness. If IV contrast administration is contraindicated, patients should have CT scan without contrast and bone scan or MRI and bone scan.
  * MRI of brain will be used for baseline assessment and tumor response assessment for CNS lesions.
  * Patients with CNS progression without systemic progression will be allowed to remain on the protocol. Local treatment, radiation, surgery, and SRS will be allowed while on protocol as deemed necessary by the treating physician.
  * Baseline imaging method(s) should be used to determine tumor response throughout course of study.
  * Measurable disease: lesions with clearly defined margins that can be accurately measured in at least one diameter (longest diameter to be recorded) with a minimum size of:

    * 10mm by CT scan (CT scan slice thickness no greater than 5mm)
    * 10mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as non-measurable)
    * 20mm by chest xray
    * Malignant lymph nodes: to be considered pathologically enlarged and measurable. Lymph node must be > 15mm in short axis when assessed by CT scan. At baseline and in follow-up, only short axis will be measured and followed.
  * Non-measurable disease: all other lesions including small lesions (longest diameter < 10mm or pathological lymph nodes with > to <15 mm (short axis), and masses with margins not clearly defined. Lesions that are considered non-measurable include:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesion
    * Lymphangitic involvement of skin or lung
* The following pre-study tests should be obtained within 14 days prior to registration in accordance with good medical practice. Results of these tests do not determine eligibility and minor deviations are acceptable if they do not impact patient safety in the judgment of the treating physician:

  * ANC > 1,000/mm3
  * platelet count > 100,000/mm3
  * hemoglobin > 9 g/dL

Exclusion Criteria:

* Patients who have received prior lapatinib for metatastic breast cancer will be excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics or psychiatric illness/social situations that would limit compliance with study requirements.
* GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (eg, Crohn's, ulcerative colitis).
* Current active hepatic or biliary disease (exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Pregnant and lactating women. Women of reproductive potential not using or unwilling to use effective birth control methods throughout the trial.
* Severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study such as:

  * Symptomatic congestive heart failure of NYHA Class III or IV
  * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C). Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA PCR testing required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
* Patients with symptomatic brain metastases who have not completed radiation therapy and/or are receiving systemic steroid therapy. Patients with leptomeningeal disease will be excluded.
* Patients with CNS progression during the trial will be allowed to receive local treatment for CNS metastases and will remain on protocol. Trial medications will be held during hte time patients are receiving radiation therapy as dictated by their treating physicians.
* Patients receiving chronic, systemic treatment with corticosteroids (of more than 4mg/day or equivalent of dexamethasone. Doses of dexamethasone of up to 8mg/day may be administered for less than 2 weeks) or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period.
* Severely impaired lung function defined as spirometry and DLCO that is < 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air.
* Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN.
* Active (acute or chronic) or uncontrolled severe infections.
* Known history of HIV seropositivity.
* Active, bleeding diathesis.
* Patients who have received prior treatment with an mTOR inhibitor (eg, sirolimus, temsirolimus, everolimus).
* Known hypersensitivity to Everolimus or other rapamycins (eg, sirolimus, temsirolimus) or to its excipients.
* Active Hepatitis B or C infection.
* Life expectancy of < 2 months.
* Prior anti-cancer therapy (eg, biologic or other targeted therapy, chemotherapy, hormonal therapy) within 2 weeks prior to Day 1 if the patient has recovered from all AEs to grade 1 except for alopecia.
* Prior investigational anti-cancer therapy within 4 weeks prior to Day 1.
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, have not recovered from side effects of any major surgery (defined as requiring general anesthesia) or may require major surgery during the course of study.
* Other malignancies within past 3 years except for adequately treated carcinoma of cervix or basal or squamous cell carcinomas of the skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-02; Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Assess the effectiveness of the combination of RAD-001 and lapatinib | 6 months
  To assess the effectiveness of the combination of RAD-001 and lapatinib as measured by the six-month Overall Response Rate in women with MBC who have progressed on trastuzumab and/or lapatinib based therapies.

SECONDARY OUTCOMES:
Overall benefit of combination | 6 months
  * Six-month Progression Free Survival.
  * Safety and Tolerability of the combination.
  * Six-month Objective CNS response rate in patients with CNS metastases.
  * Six-month Clinical benefit rate of systemic disease.
  * Six-month Clinical benefit rate in the CNS.
  * Rate of development of Brain Metastases on six months of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Qamar Khan, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Centner, Kansas City, Kansas, United States